CLINICAL TRIAL: NCT07358533
Title: Disorders Hidden Under the Guise of BMI - Metabolic Obesity in People With Normal Body Weight (MONW) - the Search for Diagnostic Markers and Its Consequences for Health
Brief Title: Metabolic Obesity in Normal Weight (MONW): Diagnostic Markers Stud
Status: Not yet recruiting | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Waldemar Pluta, Principal Investigator, Pomeranian Medical University Szczecin
Other Study IDs: Preludium 2024 - 02387
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Normal Weight Obesity; Metabolically Obese Normal Weight; Metabolic Syndrome
Keywords: Endothelial Dysfunction; Metabolic Disorders; Visceral Adiposity; Flow-Mediated Dilation; Metabolomics; Asprosin; Normal Weight
MeSH Terms: conditions — Metabolic Syndrome; Metabolic Diseases; Arachnodactyly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MONW Group: Women with normal BMI (<25 kg/m²) and excessive body fat percentage (PBF ≥ 35.78%).
- Control Group: Women with normal BMI (<25 kg/m²) and normal body fat percentage (PBF < 35.78%).

SUMMARY:
Metabolically Obese Normal Weight (MONW) represents a phenotype affecting individuals with a normal Body Mass Index (BMI) but characterized by excessive adipose tissue accumulation. This condition is associated with increased cardiovascular risk, insulin resistance, and endothelial dysfunction, yet remains underdiagnosed.

This observational longitudinal study aims to comprehensively evaluate the relationship between excessive adipose tissue deposition, endothelial dysfunction, and asprosin concentrations in young women. The study will recruit 176 healthy women aged 18-35 years with normal BMI (<25 kg/m²). Participants will be divided into two groups based on body fat percentage (PBF) assessed by dual-energy X-ray absorptiometry (DXA): the MONW group (PBF ≥ 35.78%) and the Control group (PBF < 35.78%).

The specific objectives of the study include:

* Assessment of vascular endothelial function using flow-mediated dilation (FMD) of the brachial artery.
* Evaluation of asprosin as a novel biomarker in the MONW phenotype.
* Analysis of biochemical indices including asymmetric dimethylarginine (ADMA) and von Willebrand factor (vWF).
* Advanced metabolomic profiling to identify metabolic signatures.

Participants will undergo anthropometric measurements, body composition analysis (DXA), and blood sampling for biochemical and hormonal analyses. The study aims to develop predictive models for early cardiovascular risk detection in normal-weight individuals.

DETAILED DESCRIPTION:
Study Design and Population:

This is a longitudinal observational study involving 176 healthy women aged 18-35 years. The primary aim is to identify diagnostic markers for Metabolically Obese Normal Weight (MONW) individuals. Recruitment is conducted via digital prescreening and university networks. Eligible participants must have a normal BMI (18.5-24.9 kg/m²) and stable body weight.

Group Allocation:

Participants will be divided into two groups based on Body Fat Percentage (PBF) assessed by Dual-Energy X-ray Absorptiometry (DXA):

1. MONW Group: BMI < 25 kg/m² and PBF ≥ 35.78% (threshold derived from pilot population studies).
2. Control Group: BMI < 25 kg/m² and PBF < 35.78%.

Study Procedures:

The study involves a baseline visit and a follow-up visit after 12 months.

1. Standardization: Visits are scheduled during the early follicular phase of the menstrual cycle (days 3-7) to minimize hormonal variability affecting endothelial function. Participants must fast for at least 12 hours and abstain from caffeine, smoking, and strenuous exercise for 24 hours prior.
2. Anthropometry and Body Composition: Height, weight, and circumferences (waist, hip) are measured. Whole-body composition is analyzed using DXA (Hologic QDR 4500W) to determine total and visceral fat mass.
3. Endothelial Function Assessment (FMD): Flow-mediated dilation of the brachial artery is measured using high-resolution ultrasound (Alpinion Xcube 90, linear probe L3-12). The protocol includes:

   * 1-minute baseline imaging.
   * 5-minute occlusion (cuff inflation to 250 mmHg).
   * 3-minute continuous post-occlusion imaging to assess peak diameter.
4. Biochemical Analysis: Fasting blood samples are collected for:

   * Lipid profile (TC, LDL, HDL, TG) and glucose metabolism markers (glucose, insulin, HbA1c).
   * ELISA quantification of specific biomarkers: Asprosin, Asymmetric Dimethylarginine (ADMA), von Willebrand Factor (vWF), and sex hormones (Estradiol, Testosterone, SHBG).
5. Metabolomics: Targeted and untargeted metabolomic profiling (LC-MS/MS) is performed on a subset of plasma samples to identify metabolic signatures associated with the MONW phenotype.

Data Collection:

Participants also complete standardized questionnaires regarding physical activity (IPAQ) and dietary habits (62-item FFQ-6, KomPAN). All data is pseudonymized and stored on a secured server.

ELIGIBILITY:
Inclusion Criteria:

* Written, informed consent to participate in the research.
* Gender: Female.
* Age 18-35 years.
* BMI in the range of 18.5-25 kg/m².

Exclusion Criteria:

* Thyroid disease.
* Pregnancy or breastfeeding.
* Eating disorders.
* Polycystic ovary syndrome (PCOS).
* Hormone therapy and/or use of hormonal contraceptives.
* Smoking.
* Metal or silicone implants (contraindication for DXA/body composition accuracy).
* Vitamin and/or mineral supplementation.
* Acute and/or chronic illnesses.
* Type I or II diabetes, dyslipidemia, hypertension.
* Use of hypolipemic, antihypertensive, antiglycemic, or insulin medications.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women aged 18-35 years with a normal body weight (BMI <25 kg/m²) recruited from the West Pomeranian region (Poland).
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Brachial Artery Flow-Mediated Dilation (FMD) | Baseline, 12 months
  Assessment of vascular endothelial function using high-resolution ultrasound (Alpinion Xcube 90). FMD is calculated as the percentage change in vessel diameter from baseline to peak dilation following 5-minute occlusion cuff release.

SECONDARY OUTCOMES:
Serum Asprosin Concentration | Baseline, 12 months
  Concentration of asprosin measured in serum using the ELISA method (Enzyme-Linked Immunosorbent Assay).

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar Pluta, Msc, Principal Investigator — Pomeranian Medical University in Szczecin; Anna Lubkowska, PhD, Prof., Study Director — Pomeranian Medical University in Szczecin
Locations (1):
- Pomeranian Medical University in Szczecin, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication will be shared. This includes anonymized data sets containing: anthropometric measurements (including DXA body composition), vascular endothelial function parameters (FMD), biochemical and hormonal analysis results (including asprosin, ADMA, vWF), metabolomic profiles (LC-MS/MS), and responses from dietary and physical activity questionnaires.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning at the time of publication of the associated article and will be stored for at least 10 years.
Access Criteria: Open access without restrictions. Data will be freely available to any researcher or the public for any purpose immediately upon publication.